CLINICAL TRIAL: NCT03995836
Title: Epigenetics Modifications in Morbid Obesity and Obstructive Sleep Apnea Patients (EPIMOOSA): Continous Positive Airway Pressure (CPAP) and Bariatric Surgery Impact. EPIMOOSA Study
Brief Title: Epigenetics Modifications in Morbid Obesity and Obstructive Sleep Apnea Patients: The EPIMOOSA Study
Acronym: EPIMOOSA
Status: Completed | Type: Observational
Sponsor: Aragon Institute of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 23/2014
Record Dates: First submitted 2019-05-13; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea; Morbid Obesity; Epigenetic Disorder
Keywords: Obstructive Sleep Apnea; Morbid Obesity; Epigenetics; Bariatric Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea
  Interventions: Device: CPAP; Procedure: Bariatric Surgery
- Non Obstructive Sleep Apnea
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Device: CPAP — Decision of CPAP treatment is according to clinical guidelines
  Groups: Obstructive Sleep Apnea
Procedure: Bariatric Surgery — All patients.

SUMMARY:
This study evaluates epigenetics in morbid obese patients who are waiting for bariatric surgery. A home cardiopulmonary polygraphy is performed to evaluate for the presence of sleep-disordered breathing. The principal investigator make the decision of starting CPAP among patients with obstructive sleep apnea according to current clinical guidelines. One year follow up after bariatric surgery will be performed. A total of 5 visits will be scheduled: two of them before bariatric surgery and 3 after (3, 6 and 12 months).

At every visit, all patients had: sleep questionaries, blood samples, EKG-Holter and spirometry are collected.

ELIGIBILITY:
Inclusion Criteria:

* BMI consistently > 40 kg/m2 for 3-5 years, following more than 1 year of unsuccessful controlled medical treatment
* BMI 35-40 kg/m2 with comorbidities associated with morbid obesity (MO) susceptible to improvement with weight loss (high BP, Diabetes, dyslipidemia, OSA, etc.), following more than 1 year of unsuccessful controlled medical treatment.
* A signed informed consent form

Exclusion Criteria:

* Obesity hypoventilation syndrome or treatment with positive pressure devices.
* Diagnosis of systemic inflammatory disease.
* Neoplastic diseases in the last 5 years.
* A cardiovascular event in the last 6 months.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Bariatric surgery waiting list in Royo Villanova Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Epigenetics changes in morbid obesity patient with or without obstructive sleep apnea (OSA) | 2 years
  To evaluate differences in miRNA profile among patients with morbid obesity with or without OSA Differences between exosome miRNA of MO+OSA and MO-OSA will be calculated. The results will be expressed following the method 2(delta-delta C(T)) miRNA will be analyzed: miRNA 16, 21, 34, 126, 133, 145, 146, 155, 223, 320.

SECONDARY OUTCOMES:
Impact of CPAP treatment in epigenetics changes. | 6 months
  miRNA profile will be assessed In patient with morbid obesity and coexistent OSA, at baseline and after 6 months of treatment with CPAP according with current guidelines.
Impact of weight loss due to bariatric surgery in epigenetics changes. | 12 months
  All participants included will go to bariatric surgery and 3, 6 and 12 month blood samples will be obtained.
  miRNA will be analyzed in the last 2 visits and compared with previous.

CONTACTS AND LOCATIONS:
Overall Officials: JAVIER LAZARO SIERRA, MD, Principal Investigator — Hospital Royo Villanova

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lazaro J, Sanz-Rubio D, Claveria P, Cabrejas C, Fernando J, Castanera A, Marin JM. Effect of positive pressure ventilation and bariatric surgery on extracellular vesicle microRNAs in patients with severe obesity and obstructive sleep apnea. Int J Obes (Lond). 2023 Jan;47(1):24-32. doi: 10.1038/s41366-022-01230-z. Epub 2022 Oct 25. PMID 36284205
- [Derived] Lazaro J, Claveria P, Cabrejas C, Fernando J, Daga B, Ordonez B, Segura S, Sanz-Rubio D, Marin JM. Epigenetics dysfunction in morbid obesity with or without obstructive sleep apnoea: the EPIMOOSA study. Respir Res. 2020 Feb 4;21(1):42. doi: 10.1186/s12931-020-1302-9. PMID 32019550

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03995836/Prot_SAP_000.pdf